CLINICAL TRIAL: NCT05714839
Title: A Phase 1/2 Open-label, Multicentre, Dose Escalation and Expansion Study to Investigate the Safety, Tolerability, and Clinical Activity of Belantamab as Monotherapy and in Combination With Other Treatments in Participants With Multiple Myeloma
Brief Title: A Study to Investigate the Safety and Efficacy of Belantamab for the Treatment of Multiple Myeloma When Used as Monotherapy and in Combination Treatments
Acronym: DREAMM-20
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 218670; 2022-501941-63 (EudraCT Number)
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Unconjugated belantamab antibody Belantamab Mafodotin; Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose escalation and expansion of the unconjugated belantamab antibody monotherapy (Experimental): Unconjugated belantamab antibody will be administered in participants with RRMM until progressive disease (PD)
  Interventions: Drug: Unconjugated belantamab antibody
- Part 2:Unconjugated belantamab antibody and belantamab mafodotin-given separately dose range finding (Experimental): Participants with RRMM will receive unconjugated belantamab antibody and belantamab mafodotin
  Interventions: Drug: Unconjugated belantamab antibody and belantamab mafodotin
- Part 3: Unconjugated belantamab +/- belantamab mafodotin +pomalidomide/dexamethasone in 2L+ RRMM (Experimental): Participants with second line (2L+) RRMM will receive Unconjugated belantamab antibody in combination with pomalidomide-dexamethasone backbone, with or without belantamab mafodotin.
  Interventions: Drug: Unconjugated belantamab antibody in combination with pomalidomide-dexamethasone backbone, with or without belantamab mafodotin
- Part 1b:Optional belantamab mafodotin (Experimental): Participants enrolled in Part 1 and Part 2 will be dosed until PD after which they will have the option to receive treatment with single agent belantamab mafodotin.
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Unconjugated belantamab antibody — Unconjugated belantamab antibody will be administered.
  Other Names: GSK2857914
  Arms: Part 1: Dose escalation and expansion of the unconjugated belantamab antibody monotherapy
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered.
  Other Names: GSK2857916
  Arms: Part 1b:Optional belantamab mafodotin
Drug: Unconjugated belantamab antibody and belantamab mafodotin — Unconjugated belantamab antibody and belantamab mafodotin used in combination (delivered as separate drugs) will be administered.
  Other Names: GSK2857914 and GSK2857916
  Arms: Part 2:Unconjugated belantamab antibody and belantamab mafodotin-given separately dose range finding
Drug: Unconjugated belantamab antibody in combination with pomalidomide-dexamethasone backbone, with or without belantamab mafodotin — Unconjugated belantamab antibody and belantamab mafodotin in combination with pomalidomide-dexamethasone and Unconjugated belantamab antibody in combination with pomalidomide-dexamethasone will be administered.
  Arms: Part 3: Unconjugated belantamab +/- belantamab mafodotin +pomalidomide/dexamethasone in 2L+ RRMM

SUMMARY:
The study consists of three parts:

* Part 1 The primary purpose of this part aims to evaluate the safety, tolerability, and clinical activity of escalating doses of single agent Unconjugated belantamab antibody in participants with refractory multiple myeloma (RRMM) who have received at least 3 prior therapies (4L+).
* Part 2 The primary purpose of this part is to evaluate the safety, tolerability, and clinical activity of different dose ratios of belantamab mafodotin in combination with Unconjugated belantamab antibody (delivered as separate drugs) in participants with RRMM who have received at least 3 prior therapies (4L+).
* Part 3: The Primary purpose of this part will evaluate the clinical activity of a selected dose of the unconjugated belantamab antibody, either alone or in combination with belantamab mafodotin alongside the standard of care (SoC) pomalidomide-dexamethasone backbone. The study will focus on patients with multiple myeloma who have undergone at least one prior line of therapy, including treatment with lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Participants at the time of signing the Informed Consent Form (ICF) are at least 18 years old or are of the legal age of consent in the jurisdiction in which the study is taking place.
* Participants who have histologically or cytologically confirmed diagnosis of Multiple Myeloma (MM), as defined by the international myeloma working group (IMWG) and have progressed on or following the last line of treatment Part 1 and Part 2: Participants who have received at least 3 prior lines of anti-myeloma treatments, , including lenalidomide, a proteasome inhibitor, and an anti-CD38 mAb either in combination or separately.
* Part 3: Have received at least 1 prior line of treatment anti-myeloma treatments, including lenalidomide. Prior anti-CD38-containing regimen is not mandated, however no more than 70% of participants recruited may be anti-CD38 naïve
* Participants with a history of Autologous stem cell transplant (ASCT) are eligible for study participation provided the following eligibility criteria are met:
* Transplant was greater than (>)100 days prior to screening.
* No active bacterial, viral, or fungal infection(s) present
* Eastern cooperative oncology group-performance status (ECOG-PS) of 0 to 2.
* Measurable disease defined as at least ONE of the following:
* Serum M-protein concentration greater than (>=) 0.5 gram (g)/ deciliter (dL) (>=5 gram/liter [g/L])
* Urine M-protein excretion >=200 milligram(mg)/24 hours (>=0.2 g/24 hours)
* Serum free light chain (FLC) assay: involved FLC level >=10 mg/dL (>=100 milligrams per liter [mg/L]) and an abnormal serum FLC ratio (less than [<]0.26 or >1.65)
* Have adequate organ system function as defined by the laboratory assessments
* All prior treatment-related toxicities (defined by National Cancer Institute-Common Toxicity Criteria for Adverse Events [NCI-CTCAE], v5.0, 2017) must be Grade <=1 at the time of screening except for alopecia (any grade), neuropathy (Grade <=2), or endocrinopathy managed with replacement therapy (any grade).
* Participants or legally authorized representative (LAR) capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
* Is NOT a Participant of child-bearing potential (POCBP) or
* Is a POCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency during the intervention period and for 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
* Part 3: Due to pomalidomide being a thalidomide analogue with a risk for embryofetal toxicity and prescribed under a pregnancy prevention/controlled distribution programme, POCBP will be eligible if they commit either to abstain continuously from heterosexual sexual intercourse or use two methods of reliable birth control (one method that is highly effective plus an additional barrier method), beginning at least 4 weeks prior to initiating treatment with pomalidomide, during therapy, during dose interruptions and continuing for at least 4 weeks following discontinuation of pomalidomide treatment. Thereafter, POCBP must use one contraceptive method that is highly effective (with a failure rate of less than (<)1 percentage (%) per year) for a further 3 months (total 4 months).
* The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention
* All POCBP must agree not to donate eggs (ova, oocytes) for the purpose of reproduction during this period

Exclusion Criteria:

* Diagnosis of primary Amyloid Light chain (AL) Amyloidosis, active Polyneuropathy, organomegaly, endocrinopathy, myeloma protein, and skin changes (POEMS) syndrome, primary plasma cell leukemia.
* Part 3: Active or history of venous or arterial thromboembolism within the past 3 months. Contraindications to or unwilling to undergo protocol-required anti-thrombotic prophylaxis
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent, or compliance with study procedures.
* Participant is exhibiting signs of meningeal or central nervous system involvement with MM.
* Current corneal epithelial disease except nonconfluent Superficial punctate keratitis (SPK).
* Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice.
* Presence of malignancies other than disease under study are excluded, except for any other malignancy from which the participant has been disease-free for more than 2 years and, in the opinion of the Principal investigator (PI) and GlaxoSmithKline (GSK) Medical Director, will not affect the evaluation of the effects of this clinical trial treatment on the currently targeted malignancy (MM).Participants on active surveillance or hormone treatment for non-metastatic prostate cancer are not excluded. Participants on hormone therapy for non-metastatic breast cancer are not excluded
* Evidence of cardiovascular risk including any of the following:
* Evidence of current clinically significant untreated arrhythmias, including, but not limited to, clinically significant Electrocardiogram (ECG) abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree Atrioventricular (AV) block.
* Part 1 dose escalation and Part 2 only: QT interval corrected using Fridericia's formula (QTcF) interval >480 millisecond(msec) (QT interval corrected for heart rate according to Fridericia's formula), and/or hypokalemia, and/or family history of long QT syndrome.
* Part 1 dose expansion and Part 3: Not applicable.
* History of MI, acute coronary syndromes (including unstable angina), coronary angioplasty, stenting or bypass grafting, all within three months of screening.
* Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Uncontrolled hypertension
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to Unconjugated belantamab antibody / belantamab mafodotin or any of the components of the study treatment. History of severe hypersensitivity to other Monoclonal antibodies (mAbs).
* Active infection requiring antibiotic, antiviral, or antifungal treatment.
* For serology of HBsAg+ at screen or within 3 months prior to first dose Japan only: must test hepatitis B e-antigen (HBeAg) and antibody to hepatitis B e-antigen (HBeAb.) Eligibility verification should be evaluated and agreed with a hepatologist (after they record the approval in the patient medical record).
* Known Human immunodeficiency virus (HIV) infection, unless the participant can meet specific criteria.
* Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
* Participants with Hepatitis B virus (HBV) or Hepatitis C virus (HCV) will be excluded unless specific criteria can be met.
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible.
* Part 1: Refractory to belantamab mafodotin (confirmed PD as per IMWG criteria while on belantamab mafodotin therapy or within 60 days of completing that treatment). Prior belantamab mafodotin is allowed if it was discontinued due to toxicity which subsequently resolved Note: Prior treatment with other anti-BCMA directed agents is allowed. Provided there is at least 6-month washout after the last dose of prior anti-BCMA therapy.
* Part 2: Prior belantamab mafodotin therapy is not allowed. Prior treatment with other anti-BCMA directed agents is allowed provided there is at least a 6-month washout after the last doseof prior anti-BCMA therapy to start of study therapy.
* Prior radiotherapy within 2 weeks of start of study therapy.
* Plasmapheresis within 7 days prior to the first dose of study drug.
* Prior allogeneic transplant is prohibited.
* Participants who have received prior Chimeric Antigen Receptor T-cell therapy (CAR-T) therapy with lymphodepletion with chemotherapy within 3 months of screening.
* Any major surgery (other than bone-stabilizing surgery) within 2 weeks of first dose or has not recovered fully from surgery.
* Prior treatment with a mAb within 30 days of receiving the first dose of study drugs, or treatment with an investigational agent or approved systemic anti-myeloma therapy (including systemic steroids) within 14 days or 5 half-lives of receiving the first dose of study drugs, whichever is longer.
* Part 1: Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including Granulocyte colony stimulating factor (G-CSF), Granulocyte-macrophage colony-stimulating factor (GMCSF), recombinant erythropoietin) or any thrombopoietin receptor agonists within 2 weeks before the first dose of study drug.
* Part 3:Prior Unconjugated belantamab antibody, belantamab mafodotin, and pomalidomide therapy. are not allowed. Prior treatment with other anti- B-cell maturation antigen (BCMA) directed agents is allowed provided there is at least 6-month washout after the last dose of prior anti-BCMA therapy.
* Participants must not receive live/live attenuated vaccines within 30 days prior to first dose of study treatment or whilst receiving Unconjugated belantamab antibody for at least 70 days following last study treatment.
* Known, current drug or alcohol abuse.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this trial, unless prospective Independent Review Board (IRB) approval (by chair or designee) is allowing exception to this criterion for a specific participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2029-12-03 (Estimated); Study Completion 2029-12-03 (Estimated)

PRIMARY OUTCOMES:
Part 1, 2 and 3: Number of Participants with any Adverse Event | Up to 52 months
Part 1: Number of Participants with Dose Limiting Toxicities (DLTs) | Cycle 1 (Each cycle is of 28 days)
Part 1, 2and 3: Number of Participants with Worst Case Grade Change from Baseline in Laboratory and Vital Sign Parameters | Up to 52 months
Part 1, 2 and 3: Number of Participants with severity of ocular events by the Keratopathy Visual Acuity (KVA) scale | Up to 52 months
Part 2: Overall Response Rate (ORR) | Up to 52 months
Part 3: Very Good Partial Response and better rate (VGPR+) | Up to 52 months
  VGPR+ is defined as the percentage of participants with a confirmed VGPR or better (i.e., VGPR, complete response, stringent complete response)

SECONDARY OUTCOMES:
Part 1: Observed Plasma Concentration of belantamab | Up to 52 months
Part 1: Area Under the Curve (AUC) of belantamab | Up to 52 months
Part 1: Maximum Concentration (Cmax) of belantamab | Up to 52 months
Part 1: Number of Participants with Anti-Drug Antibodies (ADA) against belantamab | Up to 52 months
Part 1: Titers of ADA against belantamab | Up to 52 months
Part 1: Overall Response Rate (ORR) | Up to 52 months
Part 2: Duration of Response (DoR) | Up to 52 months
Part 2: Observed Plasma Concentration of Total belantamab | Up to 52 months
Part 2: Area Under the Curve (AUC) of Total belantamab | Up to 52 months
Part 1: Maximum Concentration (Cmax) of Total belantamab | Up to 52 months
Part 2: Observed Plasma Concentration of belantamab mafodotin (ADC) | Up to 52 months
Part 2: Area Under the Curve (AUC) of belantamab mafodotin (ADC) | Up to 52 months
Part 2: Maximum Concentration (Cmax) of belantamab mafodotin (ADC) | Up to 52 months
Part 2: Observed Plasma Concentration of Cys-Monomethyl Auristatin-F (Cys-mcMMAF) | Up to 52 months
Part 2: Area Under the Curve (AUC) of Cys-mcMMAF | Up to 52 months
Part 2: Maximum Concentration (Cmax) of Cys-mcMMAF | Up to 52 months
Part 2: Number of Participants with ADAs against Unconjugated belantamab antibody and belantamab mafodotin | Up to 52 months
Part 2: Titers of ADAs against Unconjugated belantamab antibody and belantamab mafodotin | Up to 52 months
Part 3: Minimal residual disease (MRD) negativity rate in participants achieving at least VGPR | Up to 52 months
  MRD negativity rate is defined as the percentage of participants who achieve MRD negative status at 10-5 sensitivity threshold assessed by next generation sequencing at least once during the time of confirmed VGPR+ response per International myeloma working group (IMWG) criteria.
Part 3: Overall Response Rate (ORR) | Up to 52 months
Part 3: Duration Of Response (DoR) | Up to 52 months
Part 3: Observed Plasma Concentration of Total belantamab | Up to 52 months
Part 3: Area Under the Curve (AUC) of Total belantamab | Up to 52 months
Part 3: Observed Plasma Concentration of belantamab mafodotin (ADC) | Up to 52 months
Part 3: Area Under the Curve (AUC) of belantamab mafodotin (ADC) | Up to 52 months
Part 3: Maximum Concentration (Cmax) of belantamab mafodotin (ADC) | Up to 52 months
Part 3: Observed Plasma Concentration of Cys-Monomethyl Auristatin-F (Cys-mcMMAF) | Up to 52 months
Part 3: Area Under the Curve (AUC) of Cys-mcMMAF | Up to 52 months
Part 3: Maximum Concentration (Cmax) of Cys-mcMMAF | Up to 52 months
Part 3: Number of Participants with ADAs against Unconjugated belantamab antibody and belantamab mafodotin | Up to 52 months
Part 3: Titers of ADAs against Unconjugated belantamab antibody and belantamab mafodotin | Up to 52 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (4):
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
- Argentina (3):
  - GSK Investigational Site, Ciudadela
  - GSK Investigational Site, San Juan Bautista
  - GSK Investigational Site, Viedma
- Australia (2):
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Brazil (3):
  - GSK Investigational Site, Joinville
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Japan (4):
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Poland (2):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lublin
- GSK Investigational Site, Seoul, South Korea
- Taiwan (2):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taipei
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Kayseri
- United Kingdom (3):
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/